CLINICAL TRIAL: NCT04968145
Title: Home To Stay: a Randomized Controlled Trial Evaluating the Effect of a Post-discharge Mobile App on 30-day Re-admission Following Elective Colorectal Surgery
Brief Title: Home To Stay: a Randomized Trial Evaluating a Post-discharge Mobile App for Elective Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Division of General Surgery , Mt. Sinai Hospital (Other)
Responsible Party: Principal Investigator, Amandeep Pooni, Research Fellow, Division of General Surgery , Mt. Sinai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HomeToStay
Record Dates: First submitted 2021-07-13; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Colorectal Cancer; Inflammatory Bowel Diseases; Utilization, Health Care; Surgery; Post Discharge Monitoring
MeSH Terms: conditions — Colorectal Neoplasms; Inflammatory Bowel Diseases; Patient Acceptance of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Participants in the control group receive routine follow up care which consists of (i) written instructions regarding potential complications and the contact information of their treating surgeon, (ii) a follow up telephone call 4 weeks following discharge by a member of the health care team and (iii) an in-person follow up visit in clinic with the treating surgeon 4-6 weeks following discharge.
- Intervention Group (Experimental): The participants in the intrevention group receive the same routine care as the control group in addition to post discharge monitoring with the Home to Stay app
  Interventions: Other: Home To Stay Mobile Health Application

INTERVENTIONS:
Other: Home To Stay Mobile Health Application — Home to stay is an integrated discharge monitoring system with a mobile application. Features of the application include a "Daily Health Check" to report on post-operative recovery, picture taking capability to photograph incisions/wounds and educational information on post-operative care at home.
  Patients will complete a "Daily Health Check" on post-discharge Day #1-14, #21 and #30. The Daily Health Check consists of a series of questions specific to colorectal surgery as well as the Quality of Recovery (QoR-15) questionnaire. After completion, the participant will receive a list of recommendations tailored to their responses including relevant education modules, to contact the surgical team or in urgent cases to go to the nearest emergency room. The participants' responses will be monitored daily via a secure web site. Any participants' responses in the extreme ranges are automatically "red flagged" and notify the health care team that a follow up telephone call is required.
  Arms: Intervention Group

SUMMARY:
A single center randomized controlled trial to evaluate the effect of a post-discharge mobile health application on 30-day re-admission and patient reported outcomes following elective colorectal surgery

DETAILED DESCRIPTION:
Background: Following elective colorectal surgery, rates of re-admission are high and result in significant healthcare resource use. However, up to 20% of these re-admissions may be preventable. This represents an opportunity to improve patient outcomes, reduce health care utilization and costs through targeted interventions.

Home To Stay is an integrated discharge monitoring program using a mobile app platform that was developed to support the needs of patients following discharge after colorectal surgery. In the initial pilot testing, the 30-day re-admission rate for patients using Home to Stay was reduced from 18% to 6% and patient anxiety was reduced in over 75% of the participants.

Methods: This study is a two arm, single center, randomized control trial that will be conducted in the colorectal unit of an academic tertiary care center. Patients will be randomized1:1 using a single randomized consent design to either usual follow up in the control group or post discharge monitoring with Home to Stay in the intervention group.

Objective: The objective of this study is to evaluate the Home to Stay app and its effect on healthcare utilization and patient reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective, inpatient colorectal surgery
* Able to speak and read in English
* Able to provide informed consent
* Have access to a smartphone/tablet or desktop computer with internet access

Exclusion Criteria:

* Patients undergoing semi-elective/emergent procedure
* Patients undergoing elective day surgery
* Expected post operative admission of less than 3 days
* Discharge to another institution (rehabilitation facility/nursing home/long term care).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2020-01-21 (Actual); Study Completion 2020-01-21 (Actual)

PRIMARY OUTCOMES:
30-day re-admission | 30 Days
  Patient reported re-admission to any hospital within 30 days of discharge following surgery

SECONDARY OUTCOMES:
30-day ER visits | 30 Days
  Patient reported presentation to any hospital emergency room within 30 days of discharge following surgery
30-day primary care visits | 30 Days
  Patient reported presentation to their primary care physician within 30 days of discharge following surgery
30-day unplanned health care visits | 30 Days
  A composite of any re-admission, ER presentation or primary care visit within 30 days following the date of discharge.
Patient reported outcomes | 30 Days
  satisfaction with the discharge process, overall well-being and level of anxiety during 30-day post-discharge period were rated on a 10- point Likert scale

CONTACTS AND LOCATIONS:
Locations (1):
- Mt Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guinier D, Mantion GA, Alves A, Kwiatkowski F, Slim K, Panis Y; Association Francaise de Chirurgie. Risk factors of unplanned readmission after colorectal surgery: a prospective, multicenter study. Dis Colon Rectum. 2007 Sep;50(9):1316-23. doi: 10.1007/s10350-007-0310-x. PMID 17665252
- [Background] Li LT, Mills WL, White DL, Li A, Gutierrez AM, Berger DH, Naik AD. Causes and prevalence of unplanned readmissions after colorectal surgery: a systematic review and meta-analysis. J Am Geriatr Soc. 2013 Jul;61(7):1175-81. doi: 10.1111/jgs.12307. Epub 2013 Jun 3. PMID 23730901
- [Background] Wick EC, Shore AD, Hirose K, Ibrahim AM, Gearhart SL, Efron J, Weiner JP, Makary MA. Readmission rates and cost following colorectal surgery. Dis Colon Rectum. 2011 Dec;54(12):1475-9. doi: 10.1097/DCR.0b013e31822ff8f0. PMID 22067174
- [Background] Burke RE, Coleman EA. Interventions to decrease hospital readmissions: keys for cost-effectiveness. JAMA Intern Med. 2013 Apr 22;173(8):695-8. doi: 10.1001/jamainternmed.2013.171. PMID 23529659
- [Background] Ceppa EP, Pitt HA, Nakeeb A, Schmidt CM, Zyromski NJ, House MG, Kilbane EM, George-Minkner AN, Brand B, Lillemoe KD. Reducing Readmissions after Pancreatectomy: Limiting Complications and Coordinating the Care Continuum. J Am Coll Surg. 2015 Sep;221(3):708-16. doi: 10.1016/j.jamcollsurg.2015.05.012. Epub 2015 May 27. PMID 26228016
- [Background] Jack BW, Chetty VK, Anthony D, Greenwald JL, Sanchez GM, Johnson AE, Forsythe SR, O'Donnell JK, Paasche-Orlow MK, Manasseh C, Martin S, Culpepper L. A reengineered hospital discharge program to decrease rehospitalization: a randomized trial. Ann Intern Med. 2009 Feb 3;150(3):178-87. doi: 10.7326/0003-4819-150-3-200902030-00007. PMID 19189907
- [Background] Jones CE, Hollis RH, Wahl TS, Oriel BS, Itani KM, Morris MS, Hawn MT. Transitional care interventions and hospital readmissions in surgical populations: a systematic review. Am J Surg. 2016 Aug;212(2):327-35. doi: 10.1016/j.amjsurg.2016.04.004. Epub 2016 Jun 1. PMID 27353404
- [Background] Keng CJS, Goriawala A, Rashid S, Goldstein R, Schmocker S, Easson A, Kennedy E. Home to Stay: An Integrated Monitoring System Using a Mobile App to Support Patients at Home Following Colorectal Surgery. J Patient Exp. 2020 Dec;7(6):1241-1246. doi: 10.1177/2374373520904194. Epub 2020 Feb 12. PMID 33457571
- [Background] Sedgwick P, Hooper C. What are randomised consent designs? BMJ. 2014 Jul 25;349:g4727. doi: 10.1136/bmj.g4727. No abstract available. PMID 25063074
- [Background] Stark PA, Myles PS, Burke JA. Development and psychometric evaluation of a postoperative quality of recovery score: the QoR-15. Anesthesiology. 2013 Jun;118(6):1332-40. doi: 10.1097/ALN.0b013e318289b84b. PMID 23411725
- [Background] De La Cruz Monroy MFI, Mosahebi A. The Use of Smartphone Applications (Apps) for Enhancing Communication With Surgical Patients: A Systematic Review of the Literature. Surg Innov. 2019 Apr;26(2):244-259. doi: 10.1177/1553350618819517. Epub 2019 Jan 2. PMID 30602332
- [Background] Patel B, Thind A. Usability of Mobile Health Apps for Postoperative Care: Systematic Review. JMIR Perioper Med. 2020 Jul 20;3(2):e19099. doi: 10.2196/19099. PMID 33393925
- [Background] Jaensson M, Dahlberg K, Eriksson M, Nilsson U. Evaluation of postoperative recovery in day surgery patients using a mobile phone application: a multicentre randomized trial. Br J Anaesth. 2017 Nov 1;119(5):1030-1038. doi: 10.1093/bja/aex331. PMID 29077818
- [Background] Dahlberg K, Philipsson A, Hagberg L, Jaensson M, Halleberg-Nyman M, Nilsson U. Cost-effectiveness of a systematic e-assessed follow-up of postoperative recovery after day surgery: a multicentre randomized trial. Br J Anaesth. 2017 Nov 1;119(5):1039-1046. doi: 10.1093/bja/aex332. PMID 29077819
- [Background] Armstrong KA, Coyte PC, Brown M, Beber B, Semple JL. Effect of Home Monitoring via Mobile App on the Number of In-Person Visits Following Ambulatory Surgery: A Randomized Clinical Trial. JAMA Surg. 2017 Jul 1;152(7):622-627. doi: 10.1001/jamasurg.2017.0111. PMID 28329223